Baptist Health IRB IRB approval: 8/25/2022 Last approval: 8/25/2022 Expires: 8/24/2023 IRB#: 21-152

#### Consent for children 7-13 years old



What is a research study?

Research studies help us learn new things. We can test new ideas. First, we ask a question. Then we try to find the answer.

This paper talks about our research and the choice that you have to take part in it. We want you to ask us any questions that you have. You can ask questions any time.

### Important things to know...

- You get to decide if you want to take part.
- You can say 'No' or you can say 'Yes'.
- No one will be upset if you say 'No'.
- If you say 'Yes', you can always say 'No' later.
- You can say 'No' at any time.
- We would still take good care of you no matter what you decide.





Why are we doing this study?

We are doing this research study to find out more about the impact of an educational intervention on improving healthy lifestyle behaviors (nutrition, physical activity, screen time, and sleep).



What would happen if I join this study?

If you decide to be in this research study, we would ask you to do the following:

- Take a test: You will answer questions. The questions will be used to find out what you know and do in your daily activities (nutrition, physical activity, screen time, and sleep).
- Do something: You will be asked to join an online presentation on healthy lifestyle knowledge and behaviors with your parent(s). This will last about 45 minutes. It will be recorded and emailed 1 week after the presentation,

Baptist Health IRB IRB approval: 8/25/2022 Last approval: 8/25/2022 Expires: 8/24/2023 IRB#: 21-152



# Could bad things happen if I join this research study?

Some of the things that we will ask you to do might make you uncomfortable or be hard to do. Some of the questions or tests might be hard to answer. Answering the questionnaires and watching the educational presentation may make you tired. We will try to make sure that no bad things happen. Remember, you can skip any questions you do not want to answer/not do something if you don't want to/stop taking part at any time.



## Could the research study help me?

We think that being in this research study may help you because it can teach you how to make healthy lifestyle changes. We also hope that someday the research study will help other kids like you.



## What else do I need to know about this research study?

If you don't want to be in the study, you don't have to be. You can stop being in the study at any time. If you want to stop, please tell someone on the research team.

To thank you for being in the research study we will give you and your parent/legal guardian a \$5.00 Amazon E-Gift Card with completion of the 3 activities associated with the project: presurvey, educational presentation, and post-survey. You should talk with your parents about how you would like to use this.

You can ask questions at any time. You can talk to Rachel Sharp, BSN, RN, CPN, DNP-FNP Student, <u>rls14c@my.fsu.edu</u>. Ask us any questions you have. Take the time you need to make your choice.